CLINICAL TRIAL: NCT02776007
Title: Patients Perceptions of Using the Libre System Compared With Conventional SMBG in Adolescents With Type 1 Diabetes The Libre Sat Trial
Brief Title: Patients Perceptions of Using the "Libre" System Compared With Conventional SMBG in Adolescents With Type 1 Diabetes The Libre Sat Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMC023516Ctil
Record Dates: First submitted 2016-04-12; First posted 2016-05-18 (Estimated); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Type 1 Diabetes
Keywords: Continuous Glucose Monitoring System
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Libre Flash CGMS (Continuous Monitoring System) (Experimental): Patients will use the Libre Flash Continuous Glucose Monitoring System for 12 weeks for their glucose Management
  Interventions: Device: Libre Flash CGMS
- SMBG (Active Comparator): Patients will use Self-Monitoring of Blood Glucose for 12 weeks for their glucose management
  Interventions: Device: Self-Measurement Blood Glucose

INTERVENTIONS:
Device: Libre Flash CGMS
  Arms: Libre Flash CGMS (Continuous Monitoring System)
Device: Self-Measurement Blood Glucose — Patients will use their personal glucose meter to perform Self-Measurement Blood Glucose
  Arms: SMBG

SUMMARY:
The Libre- flash glucose monitoring system is an episodic real-time data on demand device. This means that patients can measure their glucose level when they choose by scanning the device, while at the same time a sensor automatically measures and continuously stores glucose readings day and night. Every scan shows the current glucose reading and the last 8 hours of glucose. There are no alarms and the system does not require calibration.

In the present study we aim to evaluate treatment satisfaction and comfort using the Libre flash glucose monitoring system compared to conventional Self Measurement of Blood Glucose (SMBG) in adolescents with type 1 diabetes that discontinued using continuous glucose monitoring.

The second aim of the study is to evaluate the rate of use and the impact of Libre use compared to Self-Measurement of Blood Glucose among adolescents who are sub-optimally controlled and stopped using Continuous Glucose Monitoring. The study is an investigator initiated study, single-center, randomized, parallel study of 12 weeks with an optional cross-over 12 weeks extension period .

ELIGIBILITY:
Inclusion Criteria:

* The subject has documented Type 1 Diabetes , as defined by the American Diabetes Association and World Health Organization for at least 1 year prior to study enrollment
* The subject used continuous glucose monitoring until 3 months or more before the study start
* Age 12-17 years
* The subject has an HbA1c value > 7.5% at time of screening visit
* The subject is willing to follow study instructions
* Subject is available for entire study duration

Exclusion Criteria:

* Concomitant diseases that influence metabolic control or other medical condition, which in the Investigator's opinion, may compromise patient safety
* Significant co-morbidity that, in the opinion of the investigators would preclude participation in the study
* Any significant diseases or conditions including psychiatric disorders and substance abuse that in the opinion of the investigator is likely to affect the subject's ability to complete the study or compromise patient's safety
* Subject is taking or has taken oral or parenteral glucocorticoids within 1 month prior to screening, or plans to take oral or parenteral glucocorticoids within the planned study duration. Exceptions: Short term oral or parenteral glucocorticoids up to 7 days
* Subject has known allergy to medical grade adhesives
* Subject is participating in another study of a medical device or drug that could affect glucose measurements or glucose management or receipt of any investigational medical product within 1 month prior to screening
* Female subject of child-bearing potential who have a positive pregnancy test at screening, is pregnant, breast-feeding, or planning to become pregnant within the planned study duration or is not using adequate contraceptive methods
* Subject diagnosed with current eating disorder such as anorexia or bulimia
* Subject has a history of one or more episodes of Diabetes Keto-Acidosis requiring hospitalization within a month prior to screening
* Subject has unstable or rapidly progressive renal disease or is receiving dialysis
* Subject has active proliferating retinopathy
* Subject has current or recent history of alcohol or drug abuse
* Subject has visual impairment or hearing loss, which in the Investigator's opinion, may compromise patient ability to perform study procedures safely
* Any disease or condition that may influence the HbA1C testing

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Diabetes Treatment satisfaction questionnaire | At the final visit- week 12
Libre-user evaluation questionnaire | At the final visit-week 12
  20-item questionnaire that asses treatment satisfaction with the Libre including ease of use, comfort, pain, design and system operation. The questionnaire will be scored to a final score integrating all items to a total score

SECONDARY OUTCOMES:
Glycemic control measured by HbA1c | At the final visit-week 12

OTHER OUTCOMES:
Number of blood glucose measurements at each arm | At the final visit-week 12
Number of flash glucose measurements at the intervention arm | At the final visit-week 12
Percentage of glucose sensor readings within the range of 70 to 180 mg/dl | At the final visit-week 12
Percentage of glucose sensor readings below 60 mg/dl | At the final visit-week 12
Percentage of glucose sensor readings above 240 mg/dl | At the final visit-week 12
Average of glucose sensor readings | Week 12
  Average of glucose sensor readings (per 24 hours)
Standard Deviation of glucose sensor readings | Week 12
  Standard Deviation of glucose sensor readings (per 24 hours)
  )
HbA1c change from baseline to the end of the first intervention period | At the final visit-week 12
HbA1c change from baseline to the end of the second intervention period | At the final visit-week 12
Average fasting blood glucose level | At the final visit-week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Schneider Children's Medical Center, Petah Tikva, Israel